CLINICAL TRIAL: NCT06751888
Title: Controlled CO2 Inhalation to Increase Blood Pressure in Neurogenic Orthostatic Hypotension: a Proof-of-Concept Novel Therapy Study
Brief Title: Controlled CO2 Inhalation in NOH
Acronym: CO2-nOH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: REB24-1780
Record Dates: First submitted 2024-12-20; First posted 2024-12-30 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Neurogenic Orthostatic Hypotension
Keywords: Neurogenic Orthostatic Hypotension; Autonomic; Cardiovascular; Therapies; Quality-of-life; Symptom-management; Novel

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 0% CO2 Arm (Sham Comparator): In this arm, participants will breathe with the CO2 delivery device providing no exogenous CO2 while supine and during a 10-min HUT test.
  Interventions: Device: Controlled CO2 delivery (Sham)
- Controlled CO2 Inhalation Arm (Experimental): In this arm, participants will breathe with the CO2 delivery device in the supine position until BP levels increase. Once a BP increase is observed, participants will be tilted upright and will continue to breathe with the inhalation device during a 10-min HUT test.
  Interventions: Other: Controlled CO2 delivery

INTERVENTIONS:
Other: Controlled CO2 delivery — The use of a controlled CO2 delivery offers a straightforward way to increase arterial CO2. Controlled CO2 inhalation may offer a novel hemodynamic therapy for patients with Neurogenic Orthostatic Hypotension
  Arms: Controlled CO2 Inhalation Arm
Device: Controlled CO2 delivery (Sham) — For this intervention, we will be using this device set at 0% CO2 for our sham comparison.
  Arms: 0% CO2 Arm

SUMMARY:
This study focuses on neurogenic orthostatic hypotension (nOH), which is a disorder characterized by an abnormal drop in blood pressure (BP) within 3-minutes of standing. Patients with nOH experience debilitating symptoms including light-headedness, falls, and fainting. Patients often struggle with day-to-day tasks that require standing, with a reduced quality-of-life. Current therapies for nOH have limited effectiveness and unwanted side effects. Our lab has found that raising blood CO2 levels (hypercapnia) in the lab increases BP when standing in patients with nOH. We now aim to test the CarboHaler, an exogenous controlled CO2 delivery device, in this study to see if increasing CO2 levels through controlled CO2 inhalation can improve BP and reduce symptoms in patients with nOH when standing up. On the study day, participants will undergo two Head-up Tilt (HUT; upright) tests with different breathing protocols: one with and one without exogenous CO2 delivery provided by a CO2 inhalational device. We will record heart rate, blood pressure, and breathing parameters. We will also assess upright symptoms using the Vanderbilt Orthostatic Symptoms Score. Our primary outcome is the magnitude of the change in systolic BP from lying down to standing, which will be compared with and without exogenous CO2 delivery. We hypothesize that exogenous CO2 delivery provided by a CO2 inhalational device will raise CO2 enough to increase standing BP, which could reduce the debilitating symptoms experienced by patients with nOH. We hope that these data will support future clinical trials, with the long-term goal of creating a simple, low-cost treatment for increasing quality-of-life for patients with nOH.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Male and Female
* Physician diagnosis of Neurogenic Orthostatic Hypotension
* Non-smokers.
* Able and willing to provide informed consent.
* Ability to travel to Libin Cardiovascular Institute Autonomic Testing Lab at the University of Calgary, Calgary, AB.

Exclusion Criteria:

* Pregnant or breast-feeding females
* Subjects with chronic heart failure or severe pulmonary disease who are unable to climb one flight of stairs due to shortness of breath.
* Presence of failure of other organ systems or systemic illness that can affect autonomic function or the participant's ability to cooperate. These include dementia, alcohol and/or drug abuse.
* Other factors which in the investigator's opinion would prevent the participant from completing the protocol, including poor compliance during previous studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Magnitude of the systolic blood pressure (SBP) response | Start of in-lab study day to the end of the in-lab study day
  The primary outcome measures will be the magnitude of the systolic blood pressure (SBP) response (ΔSBP = Head Up Tilt - Supine) during 0% CO2 vs. Controlled CO2 inhalation.

SECONDARY OUTCOMES:
Change in Cerebral Blood Flow (ΔCBFv) | Start of in-lab study day to the end of the in-lab study day
  Secondary outcome measures will be the change in Cerebral Blood Flow (ΔCBFv) for each arm of the study.
Change in Vanderbilt Orthostatic Symptom Scores (ΔVOSS) | Start of in-lab study day to the end of the in-lab study day
  Secondary outcome measures will be the change in Vanderbilt Orthostatic Symptom Scores (ΔVOSS) for each arm of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No